CLINICAL TRIAL: NCT05066607
Title: A Phase 2, Open Label, Multicenter, Single-stage Study to Evaluate the Efficacy of Isatuximab Plus Pomalidomide and Dexamethasone (IPd), in Patients With AL Amyloidosis Not in VGPR or Better After Any Previous Therapy
Brief Title: Isatuximab Plus Pomalidomide and Dexamethasone Association for Patients With AL Amyloidosis Not in VGPR or Better After Any Previous Therapy
Acronym: IsAMYP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone du Myelome (Network)
Collaborators: Sanofi (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFM 2020-01
Record Dates: First submitted 2021-08-24; First posted 2021-10-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: AL Amyloidosis
Keywords: Amyloidosis; Isatuximab; Pomalidomide; Dexamethasone; Not in VGPR; Not in first line of treatment
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — isatuximab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-stage (Experimental): Patient eligible to enter the study will receive 9 to 12 cycles (according to response) of intravenous Isatuximab (10 mg/kg) and oral Pomalidomide 4 mg from day 1 to day 21 and Dexamethasone 10-20 mg weekly on days 1, 8, 15 and 22.
  Each cycle will be of 28 days duration. During cycle 1, Isatuximab will be administered weekly on days 1, 8, 15, and 22 then days 1 and 15 in subsequent cycles from cycle 2 to 9 or 12.
  For each individual patient, the treatment period will be 12 months, unless CR at the completion of 9 cycles, disease progression or unacceptable toxicity occurs. The duration of follow-up for overall survival will be 1 year after the last patient enters overall survival follow-up.
  Interventions: Drug: Isatuximab

INTERVENTIONS:
Drug: Isatuximab — Patient will receive the association of Isatuximab, Pomalidomide and Dexamethasone during 9 or 12 cycles.
  Other Names: Pomalidomide; Dexamethasone

SUMMARY:
This phase 2 study ain to evaluate the efficacy of Isatuximab plus Pomalidomide and Dexamethasone (IPd), in patients with AL amyloidosis not in VGPR or better after any previous therapy. It will enrolled 46 patients (34 in France and 12 in Australia) through 15 sites (11 in France and 4 in Australia).

DETAILED DESCRIPTION:
Systemic AL amyloidosis is a rare disease caused by the deposition of misfolded monoclonal immunoglobulin free light chains (FLC) in various tissues and organs. It is usually associated with a clonal plasma cell dyscrasia with a low tumor burden. Treatment of AL amyloidosis relies mainly on chemotherapy aimed at suppressing the underlying plasma cell clone secreting monoclonal FLC.

The organ responses and the survival are greatly influenced by the degree of hematological response evaluated by the decrease in serum FLC that has been the principal endpoint in recent trials in AL amyloidosis. The goal of treatment is to reach at least a very good partial response (VGPR) defined as a difference between the involved FLC and the normal one below 40 mg/L.

Over the last 5 years, monoclonal antibodies (mAb) as daratumumab and Isatuximab (anti CD38 mAb) has emerged as a breakthrough targeted therapies for patients with multiple myeloma (MM).

CD38, is a type II transmembrane glycoprotein that functions both as a signal-transducing receptor and a multifunctional ectoenzyme. The expression of CD38 is increased in MM and AL amyloidosis plasma cells.

Daratumumab (DARA) is an IgG 1k human mAb that received initial approval as monotherapy in patients with heavily pretreated RRMM and who were refractory to proteasome inhibitors (PIs) and immunomodulatory drugs (IMiD®). DARA has since been approved in combination with Lenalidomide/Dexamethasone1,2 and Bortezomib/Dexamethasone3,4 for the treatment of frontline and relapsed/refractory (RR) MM patients.

IFM and other groups previously demonstrated that DARA in monotherapy is safe and effective in relapsed AL amyloidosis patients5. Our prospective phase II study showed that about 70 to 80% of patients have a response but only around 50% reached a VGPR.

DARA activity could be increased with IMiD® as treating plasma cells with IMiD®, such as pomalidomide or lenalidomide, has been shown to increase the expression of CD38 levels on the surface of these cells.

In AL amyloidosis, the Italian and the British groups demonstrated that pomalidomide is very effective and better tolerated than lenalidomide especially in patients with renal insufficiency6,7. The dose of pomalidomide (4 mg) was like the dose used in MM.

Combining an anti CD38 mAb to pomalidomide could therefore be an attractive regimen for relapsed AL amyloidosis patients.

Isatuximab (ISA) is another IgG1 κ mAb that binds selectively to a unique epitope on the human CD38 receptor and has anti plasma cells activity via multiple mechanisms of action. In a previous phase 1b study, around 65% of patients with relapsed and refractory multiple myeloma achieved an overall response with a combination of Isatuximab with Pomalidomide and low-dose Dexamethasone.

The addition of Isatuximab to Pomalidomide-Dexamethasone was used in a large phase III study in RRMM8. Safety profile was also favorable, and these results granted an approval of the combination of ISA plus Pomalidomide (4 mg) and Dexamethasone in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Histologic diagnosis of AL amyloidosis;
3. Patients should have received at least one line with an alkylating agent and/or a PI, and Dexamethasone and not be in VGPR (or better) at the time of inclusion (patients who did not reach VGPR before, or patients in VGPR or better before but with a hematological relapse at the time of inclusion can be included);
4. Measurable hematologic disease: difference between involved and uninvolved FLC > 50 mg/L with an abnormal k/l ratio;
5. Symptomatic organ involvement (heart, kidney, liver/GI tract, peripheral nervous system) (See Appendix 1);
6. Wash-out period of at least 4 weeks from previous antitumor therapy or any investigational treatment or 5 half-lives from previous antibodies, whichever is longer.
7. Adequate bone marrow function prior to 1st drug intake (C1D1), without transfusion or growth factor support within 5 days prior to 1st drug intake, defined as:

   * Absolute neutrophils count ≥ 1000/mm3,
   * Platelets ≥ 75000/mm3,
   * Hemoglobin ≥ 8.0 g/dL,
8. Adequate organ function defined as:

   * Serum ASAT or ALAT ≤ 3.0 X Upper Limit of the normal range (ULN),
   * Serum total bilirubin level < 1.5 x ULN, unless for subjects with Gilbert's syndrome where the direct bilirubin should then be ≤ 2.0 x ULN.
9. ECOG status ≤ 2
10. Male participants must agree to use contraception during the intervention period and for at least 5 months after the last dose of IsaPd and refrain from donating sperm during this period.

    * Female participants are eligible to participate if they are not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a Female of childbearing potential (FCBP), OR a FCBP who must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting study medication and before each cycle of study treatment and must either commit to continue abstinence from heterosexual intercourse or apply a highly effective method of birth control 4 weeks before initiation of treatment, during the intervention period and for at least 5 months after IsaPd treatment,
    * Female patients who are postmenopausal for at least 1 year before the screening visit, or are surgically sterile, or if they are of childbearing potential, agree to practice effective methods of contraception from the time of signing the informed consent through 30 days after the last dose of study drug, or agree to completely abstain from intercourse (serum pregnancy test must be performed for all women of childbearing potential at the beginning of each cycle during the study. In addition, a pregnancy test may be done at any time during the study at the discretion of the investigator if a subject misses a period or has unusual menstrual bleeding);
11. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Presence of non-AL amyloidosis
2. AL amyloidosis with isolated soft tissue involvement
3. Bone marrow plasma cells >30% and clinically symptomatic multiple myeloma with lytic bone lesions
4. NT-proBNP > 8500 ng/L and hs-troponin I > 100 ng/L or hs-troponin T > 50 ng/L (cardiac stage IIIb patients)
5. Repetitive ventricular arrhythmias on 24h Holter ECG despite anti-arrhythmic treatment sustained ventricular tachycardia, aborted ventricular fibrillation, atrioventricular nodal or sinoatrial nodal dysfunction with no pacemaker
6. Chronic atrial fibrillation with uncontrolled heart rate
7. Significant cardiac dysfunction; myocardial infarction within 12 months; unstable poorly controlled angina pectoris
8. Uncorrected valvular disease unrelated to AL amyloid cardiomyopathy
9. QT interval as corrected by Fridericia's formula >550 msec without pacemaker,
10. Undergoing dialysis
11. Ongoing toxicity (excluding alopecia and those listed in eligibility criteria) from any prior therapy >G1 (NCI-CTCAE v5.0)
12. Supine systolic blood pressure <90 mm Hg, or symptomatic orthostatic hypotension, defined as a decrease in systolic blood pressure upon standing of <80 mmHg despite medical management (i.e. midodrine, fludrocortisones) in the absence of volume depletion
13. Previous anti-CD38 therapy or Pomalidomide therapy (if refractory to Pomalidomide)
14. Hypersensitivity to IMiD® defined as any hypersensitivity reaction leading to stop IMiD® within the 2 first cycles or toxicity, which does meet intolerance definition
15. Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, polysorbate 80, poloxamer 188, sucrose or any of the other components of study treatment that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents
16. History of malignancy (other than AL amyloidosis) within 3 years before the date of inclusion (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years)
17. Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results
18. Active systemic infection and severe infections requiring treatment with a parenteral administration of antibiotics
19. Received any investigational drug within 14 days or 5 half-lives of the investigational drug prior to initiation of study intervention, whichever is longer. In case of very aggressive disease (i.e acute leukemia) delay could be shortened after agreement between sponsor and investigator, in absence of residual toxicities from previous therapy
20. Known positive for HIV or active hepatitis A, B or C:

    * Uncontrolled or active HBV infection: Patients with positive HBsAg and/or HBV DNA

    Of note:

    Patient can be eligible if anti-HBc IgG positive (with or without positive anti-HBs) but HBsAg and HBV DNA are negative.
    * If anti-HBV therapy in relation with prior infection was started before initiation of IMP, the anti-HBV therapy and monitoring should continue throughout the study treatment period.

    Patients with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative and all the other study criteria are still met.
    * Active HCV infection: positive HCV RNA and negative anti-HCV.

    Of note:

    Patients with antiviral therapy for HCV started before initiation of IMP and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.

    Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible
21. Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Hematologic Response | At the end of Cycle 6 (each cycle is 28 days)
  To assess hematologic response (VGPR or better i.e. dFLC < 40 mg/L, CR including modified CR*, low-dFLC response (dFLC < 10 mg/L), iFLC < 10 mg/l) achieved after 6 cycles of Isa-Pd.
  *: If iFLC <ULN and serum and urine immunofixation are negative, then neither a normal uFLC level nor a normal FLC ratio are required for complete response (CR).

SECONDARY OUTCOMES:
Overall Hematologic Response Rate | At the completion of the 1st, 2nd, 4th, 6th, 9th and 12th cycles (each cycle is 28 days)
  To assess in all patients according to their disease history Overall Hematologic Response Rate (VGPR, CR, modified CR*, Low-dFLC response (dFLC < 10 mg/L), iFLC < 10 mg/l and PR) at the completion of the 1st, 2nd, 4th, 6th, 9th and 12th cycles.
  *: If iFLC <ULN and serum and urine immunofixation are negative, then neither a normal uFLC level nor a normal FLC ratio are required for complete response (CR).
Efficacy Measurement: Progression-free survival (PFS) | During the intervention and at 1 year
  Time from the inclusion to either progressive disease or death
Efficacy Measurement: relapse-free survival (RFS) | During the intervention
  To evaluate the relapse-free survival (RFS)
Efficacy Measurement: Organ response rate (OrRR) | 1 year
  To evaluate the Organ response rate at 1 year
Efficacy Measurement: Overall Survival (OS) | Though study completion, an average of 33 months
  Time from initial inclusion to death
Time to and the duration of haematologic and organ responses | During the intervention
  To evaluate the time to and the duration of haematologic and organ responses
Safety analysis | Until 30 days post last dose of protocol treatment
  Rate of adverse events that occured during treatment period
Cytogenetic: incidence of genetic translocation t(11;14) and impact on hematologic and organ response | Though study completion, an average of 33 months
  To assess the impact of t(11.14) determined by Fluorescence In Situ Hybridation (FISH) at inclusion on treatment response.
Cardiac function | After 6 cycles of IsaPd and at 1 year from start of therapy or 12 cycles of IsaPd (each cycle is 28 days).
  To assess the concentration of NT-proBNP level and evaluate the impact of the NT-proBNP level on the strain change.
Renal function | After 6 cycles of IsaPd and at 1 year from start of therapy or 12 cycles of IsaPd (each cycle is 28 days)
  To assess albumin level to proteinuria/eGFR.
Quality of Life : European Quality of Life 5 dimensions (EQ-5D-3L) | up to 15 months
  patient reported outcome to assess health status in patients. The EQ-5D (European Quality of Life 3 dimensions) measures a wide range of health conditions and treatments; it is composed of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and a visual analogue scale that records the patient's self-rated overall health state.
  Respondents rate each of these 5 dimensions from "no problem", "some problem" or "extreme problem".
  The EQ-VAS records the respondents' self-related health on a vertical, visual analogue scale. The range for EQ-VAS is from 0 (the worst health you can imagine) to 100 (=the best healt you can imagine).

OTHER OUTCOMES:
Minimal Residual Disease (MRD) | At the completion of 6 cycles of therapy or at 1 year from start of therapy (each cycle is 28 days)
  To assess Minimal Residual Disease (MRD) by NGS in bone marrow and blood at the completion of 6 cycles of therapy or at 1 year from start of therapy for patients in CR/modified CR* or low dFLC or normal iFLC (iFLC< 10 mg/L) and by Mass Spectrometry in the blood.
  *: If iFLC <ULN and serum and urine immunofixation are negative, then neither a normal uFLC level nor a normal FLC ratio are required for complete response (CR).

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud JACCARD, Pr, Principal Investigator — CHU Limoges
Locations (15):
- France (15):
  - CHU Amiens-Picardie, Amiens
  - CHRU - Hôpital du Bocage, Angers
  - CHU Caen - Côte de Nacre, Caen
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHRU Hôpital Claude Huriez, Lille
  - Centre Hospitalier Universitaire (CHU) de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Hopital Saint Eloi - CHU Montpellier, Montpellier
  - CHRU Nancy - Hôpitaux de Brabois, Nancy
  - CHRU Hôtel Dieu, Nantes
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Hôpital Saint Louis, Paris
  - CHU Poitiers - Pôle régional de Cancérologie, Poitiers
  - CHRU Hôpital de Pontchaillou, Rennes
  - Pôle IUCT Oncopole CHU, Toulouse